CLINICAL TRIAL: NCT06946498
Title: Local Anesthesia Thoracoscopy as a First Line Approach in the Diagnosis of Suspected Malignant Pleural Effusion: FLAT Trial.
Brief Title: First Local Anaesthesia Thoracoscopy for Pleural Effusion Diagnosis.
Acronym: FLAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Collaborators: Sotiria Thoracic Diseases Hospital of Athens (Other)
Responsible Party: Principal Investigator, Stratakos Grigorios, Professor of Interventional Pulmonology, National and Kapodistrian University of Athens
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: FLAT1STIPNKUA
Record Dates: First submitted 2025-04-10; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Suspected Malignant Lung Neoplasm; Pleural Effusion; Pleural Effusion, Malignant; Mesothelioma, Malignant
Keywords: Malignant Pleural Effusion; Local Anesthesia Thoracoscopy; Medical Thoracoscopy; Lung cancer; Mesothelioma; Lymphocytic Exudate
MeSH Terms: conditions — Pleural Effusion; Pleural Effusion, Malignant; Mesothelioma, Malignant; Lung Neoplasms; Mesothelioma | interventions — Thoracoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LAT Group (Experimental): The study group includes patients in whom the investigation of pleural effusion begins directly with pleural biopsy by Local Anesthesia Thoracoscopy (LAT) under conscious sedation. In these patients, imaging with chest CT and/or thoracic ultrasound has been performed and lymphocytic exudate is confirmed in fluid aspiration.
  Interventions: Procedure: Local Anesthesia Thoracoscopy; Device: Pleuroscopy with Rigid Thoracoscope and Forceps biopsies
- Control Group (No Intervention): The Control Group includes patients admitted with undiagnosed pleural lymphocytic exudate, who undergo Standard of Care (SOC) diagnostic strategies according to BTS guideline including among others, 3 samples for cytological examination (40-60 ml each), chest tube drainage, microbiological and immunological studies. If the diagnosis is not established and there is still indication for pleural biopsy patients are referred either for surgical biopsy or LAT.

INTERVENTIONS:
Procedure: Local Anesthesia Thoracoscopy — The patient is placed in a lateral decubitus, with the affected hemithorax upwards. Ensuring a venous line and full monitoring of vital functions. Mild sedation is given and a dose of Ceftriaxone is given 30 minutes before. Local anesthesia is injected in layers, starting from the skin and working up to the intercostal muscles, intercostal nerve, and periosteum of the rib.
  Development of pneumothorax is done using a 16-gauge Boutin needle. 15 spontaneous breaths are sufficient to create a pneumothorax, and entry of rigid thoracoscope into the hemithorax through a 11-13 mm Trocar. Multiple biopsies from the parietal pleura are taken and pleurodesis is made according to operator judgment. A chest drain 20-22 G is placed and sutured.
  A chest X-ray is performed 2-8 hours later after the patient is transferred to the ward. Chest drain is removed after 24h if fluid production is <250ml and lung re-expansion.
  Arms: LAT Group
Device: Pleuroscopy with Rigid Thoracoscope and Forceps biopsies — A video thoracoscope with an external light source, outer diameter 10 mm (Karl Storz), is inserted into the pleural cavity through a uniportal incision (1 - 1.5 cm) and complete inspection of the pleural cavity is performed. Parietal pleural biopsies are taken with a rigid 40 mm forceps (Karl Storz).
  Arms: LAT Group

SUMMARY:
Non randomized study with two groups. The study group includes patients with suspected malignant pleural effusion, in whom the investigation of pleural effusion begins directly with pleural biopsy by Local Anesthesia Thoracoscopy (LAT).

The Control Group includes patients who come to the same hospital and are treated with the Standard of Care (SOC) strategies were used. Efficacy of LAT, Sensitivity, Hospitalization, time to diagnosis and general safety and comfort of the groups' subjects will be assessed.

DETAILED DESCRIPTION:
Diagnostic approach of patients with with unexplained lymphocytic exudate is the main subject of the study. Minimally invasive techniques (single entry thoracoscopy with local anesthesia -LAT) have been developed for the definitive biopsy of the parietal pleura, with which, in addition to the diagnosis, a therapeutic pleurodesis can be performed at the same time. Usually, diagnostic LAT is performed only after 3 negative pleural fluid cytological tests have been performed, thus delaying the diagnostic access and treatment of the patient.

The aim of this study is to evaluate the conventional diagnostic approach used in daily clinical practice (3 consecutive punctures of pleural effusion with cytological examination and in case of insufficient diagnosis pleural biopsy, either LAT or VATS depending on the clinical assessment of the patient) with the simplest immediate performance of LAT as soon as a pleural effusion suspected of malignancy is detected. Thus two subject groups will be compared. The first (LAT Group) will undergo Local Anesthesia Thoracoscopy as the first line option for the diagnosis of the suspected MPE. The control group will undergo the standard of care recommended guidelines for the diagnosis of MPE.

ELIGIBILITY:
Inclusion Criteria:

* Undiagnosed pleural effusion with the character of a lymphocytic exudate

Exclusion Criteria:

* Empyema
* Transudate pleural effusion.
* Central airway obstruction by tumor.
* Existence of extensive adhesions that do not allow the development of iatrogenic pneumothorax and the safe entry of the thoracoscope.
* Uncontrollable cough.
* Acute respiratory failure and/or Hypercapnia.
* Performance Status: 5

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-05-23 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to Diagnosis | From enrollment to final diagnosis of MDT, assesed up to 12 months
  Time to diagnosis is defined as the period between the first thoracentesis ,showing a lymphocytic exudate, of a newly discovered pleural effusion in a patient without prior signs of pleural disease to the time of multi-disciplinary team final diagnosis involving a pathology report of biopsy samples.
Hospitalization time | From enrollment to hospital discharge, assesed up to 3 months
  The time from the patient's admission in the hospital with diagnosis of unexplained lymphocytic pleural effusion until discharge with or without final diagnosis.

SECONDARY OUTCOMES:
Patient's discomfort/pain | Day 1: immediately post-procedure. Day 2: 24hours post-procedure. Day 3 up to Day of tube removal: Every 24 hours. Time frame ends on removal of chest tube or patient dishcarge, assesment up to 2 weeks
  A Visual Analogue Scale (VAS) measures the intensity of pain the patient feels after the intervention (Medical Thoracoscopy vs Surgical Biopsy). A horizontal line ranging from 0 to 10, (0=No pain, 10=Extreme pain), is used. The patient is examined every day, until his discharge and is asked to mark on the line his respective level of discomfort/pain.
Complications | Day 1: immediately post-procedure. Day 2: 24hours post-procedure. Day 3 up to Day of tube removal: Every 24 hours. Time frame ends on removal of chest tube or patient dishcarge, assesment up to 3 months.
  We compare the rate of post interventional complications across the two groups (Surgical biopsy vs LAT)
Rate of Non Specific Pleuritis | Assesment up to 12 months
  We aim to asses wheter the rate of positive pleural biopsies for non specific pleuritis differed significantly between Surgical biopsy group and LAT group.

CONTACTS AND LOCATIONS:
Overall Officials: Grigorios Stratakos, Professor, Study Director — National and Kapodistrian University of Athens
Locations (1):
- Sotiria General Hospital of Thoracic Diseases, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No
This is a preliminary study design and for confidentiality rationales in order to protect the novelty of diagnostic strategies implemented in this research .

REFERENCES:
- [Background] Ferguson J, Tsim S, Kelly C, Alexander L, Shad S, Neilly M, Tate M, Zahra B, Saleh M, Cowell G, Banks E, Grundy S, Corcoran J, Downer N, Stanton A, Evison M, Rahman NM, Maskell N, Blyth KG. Staging by Thoracoscopy in potentially radically treatable Lung Cancer associated with Minimal Pleural Effusion (STRATIFY): protocol of a prospective, multicentre, observational study. BMJ Open Respir Res. 2023 Nov 23;10(1):e001771. doi: 10.1136/bmjresp-2023-001771. PMID 37996118
- [Background] Wan YY, Zhai CC, Lin XS, Yao ZH, Liu QH, Zhu L, Li DZ, Li XL, Wang N, Lin DJ. Safety and complications of medical thoracoscopy in the management of pleural diseases. BMC Pulm Med. 2019 Jul 10;19(1):125. doi: 10.1186/s12890-019-0888-5. PMID 31291926
- [Background] Shaikh F, Lentz RJ, Feller-Kopman D, Maldonado F. Medical thoracoscopy in the diagnosis of pleural disease: a guide for the clinician. Expert Rev Respir Med. 2020 Oct;14(10):987-1000. doi: 10.1080/17476348.2020.1788940. Epub 2020 Jul 12. PMID 32588676
- [Background] Gong L, Huang G, Huang Y, Liu D, Tang X. Medical Thoracoscopy for the Management of Exudative Pleural Effusion: A Retrospective Study. Risk Manag Healthc Policy. 2020 Dec 4;13:2845-2855. doi: 10.2147/RMHP.S287758. eCollection 2020. PMID 33324122
- [Background] Murthy V, Bessich JL. Medical thoracoscopy and its evolving role in the diagnosis and treatment of pleural disease. J Thorac Dis. 2017 Sep;9(Suppl 10):S1011-S1021. doi: 10.21037/jtd.2017.06.37. PMID 29214061
- [Background] Xu LL, Yang Y, Wang Z, Wang XJ, Tong ZH, Shi HZ. Malignant pleural mesothelioma: diagnostic value of medical thoracoscopy and long-term prognostic analysis. BMC Pulm Med. 2018 Apr 3;18(1):56. doi: 10.1186/s12890-018-0619-3. PMID 29615010
- [Background] Li D, Jackson K, Panchal R, Aujayeb A. Local Anaesthetic Thoracoscopy for Pleural Effusion-A Narrative Review. Healthcare (Basel). 2022 Oct 9;10(10):1978. doi: 10.3390/healthcare10101978. PMID 36292425
- [Background] Arnold DT, De Fonseka D, Perry S, Morley A, Harvey JE, Medford A, Brett M, Maskell NA. Investigating unilateral pleural effusions: the role of cytology. Eur Respir J. 2018 Nov 8;52(5):1801254. doi: 10.1183/13993003.01254-2018. Print 2018 Nov. PMID 30262573
- [Background] Kiani A, Abedini A, Karimi M, Samadi K, Sheikhy K, Farzanegan B, Pour Abdollah M, Jamaati H, Jabardarjani HR, Masjedi MR. Diagnostic Yield of Medical Thoracoscopy in Undiagnosed Pleural Effusion. Tanaffos. 2015;14(4):227-31. PMID 27114723
- [Background] Wu YB, Xu LL, Wang XJ, Wang Z, Zhang J, Tong ZH, Shi HZ. Diagnostic value of medical thoracoscopy in malignant pleural effusion. BMC Pulm Med. 2017 Aug 4;17(1):109. doi: 10.1186/s12890-017-0451-1. PMID 28778184
- [Background] Kassirian S, Hinton SN, Cuninghame S, Chaudhary R, Iansavitchene A, Amjadi K, Dhaliwal I, Zeman-Pocrnich C, Mitchell MA. Diagnostic sensitivity of pleural fluid cytology in malignant pleural effusions: systematic review and meta-analysis. Thorax. 2023 Jan;78(1):32-40. doi: 10.1136/thoraxjnl-2021-217959. Epub 2022 Feb 2. PMID 35110369
- [Background] Tsim S, Paterson S, Cartwright D, Fong CJ, Alexander L, Kelly C, Holme J, Evison M, Blyth KG. Baseline predictors of negative and incomplete pleural cytology in patients with suspected pleural malignancy - Data supporting 'Direct to LAT' in selected groups. Lung Cancer. 2019 Jul;133:123-129. doi: 10.1016/j.lungcan.2019.05.017. Epub 2019 May 16. PMID 31200818